CLINICAL TRIAL: NCT04271215
Title: Overweight and Obesity as Prognostic Factors for Survival in Children With Acute Lymphoblastic Leukemia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Juan Manuel Mejía Aranguré, Head of the Research Linkage Area, Coordinación de Investigación en Salud, Mexico
Other Study IDs: R-2015-785-070
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Leukemia, Lymphoblastic
Keywords: Overweight; Obesity; Survival; Children
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overweight/Obesity: BMI at diagnosis will be used. Using WHO software (version 3.2.2, World Health Organization, Geneva), the BMI-for-age Z-scores were calculated for each patient. According to WHO classification, patients were categorized as normal (- 1.9999 to 0.9999), wasted (- 2 to - 2.9999), severely wasted (≥ - 3), at risk of overweight (1-1.9999), overweight (2 to 2.9999) and obesity (≥3). In addition, the BMI percentiles cutoffs provided by CDC were: normal (p5-84.9999), underweight (< p5), overweight (p85-94.9999), and obese (≥ p95). The nutritional classification and measurements regarding weight and height recorded in clinical files will be used to classify patients' nutritional status in present research has been previously described.
  Interventions: Other: Chemotherapy protocol used

INTERVENTIONS:
Other: Chemotherapy protocol used — Chemotherapy protocol used in each participating hospital

SUMMARY:
Background: Mexico City has one of the highest incidences and mortality rates of acute lymphoblastic leukemia (ALL) in the world and a high frequency of early relapses (17%) and early mortality (15%). Otherwise, childhood overweight and obesity are reaching epidemic proportions. They have been associated with poor outcomes in children with ALL. The aim of present study is to identify if overweight and obesity are prognostic factors associated with survival rates in Mexican children with ALL. Methods: Multicenter cohort study. ALL children younger than 15 years old are included and followed-up. Overweight and obesity are classified according World Health Organization (WHO) and Centers for Disease Control and Prevention (CDC) criteria. Deaths and relapses are the main outcomes.

DETAILED DESCRIPTION:
Data collection Information regarding sex, age at diagnosis, place of residence, white blood cell (WBC) count, immunophenotype (B or T lineage), weight and height (length when appropriate) at diagnosis, and chemotherapy protocol is collected from the patients' clinical charts by previously standardized staff. Overcrowding was used as a proxy for socioeconomic status (SES) according to the Bronfman's criteria (high SES, up to 1.5 people per room; medium-low SES, more than 1.6 people per room). The risk classification is according to the criteria of the National Cancer Institute (NCI): standard risk [ages from 1 to 9.99 years; WBC count < 50 × 109/L] or as high risk [age < 1 or ≥ 10 years or WBC ≥ 50 × 109/L].

Assessment of nutritional status at diagnosis of ALL BMI at diagnosis will be used.. Using WHO software (version 3.2.2, World Health Organization, Geneva), the BMI-for-age Z-scores were calculated for each patient. According to WHO classification, patients were categorized as normal (- 1.9999 to 0.9999), wasted (- 2 to - 2.9999), severely wasted (≥ - 3), at risk of overweight (1-1.9999), overweight (2 to 2.9999) and obesity (≥3). In addition, the BMI percentiles cutoffs provided by CDC were: normal (p5-84.9999), underweight (< p5), overweight (p85-94.9999), and obese (≥ p95). The nutritional classification and measurements validation regarding weight and height recorded in clinical files used to classify patients' nutritional status in present research has been previously described. Underweight patients were excluded from the analyses.

Sample size The sample size calculation was performed using Epi-Info version 7 software taking into account a mortality outcome frequency of 10.8% in the unexposed group (normal weight patients) and a death outcome frequency of 24% for the exposed (obese/overweight patients), a statistical power of 80% and a confidence of 95%; resulting in a total "n" of 350 overweight/obese patients to be compared with the rest of the cohort that are not overweight and obese.

Statistical analysis Descriptive statistics and relative risks (RR) calculation with 95% confidence intervals (CI) will be carried out. Kaplan-Meier survival analysis will be conducted. Log-rank test will be calculated. The analyses will be conducted independently for disease-free-survival (DFS) or overall survival (OS), adjusting for variables whose effects on the studied outcomes have been previously documented (age, sex, socioeconomic status, immunophenotype, NCI risk classification, and chemotherapy protocol). A Cox proportional hazard model will be used. Hazard ratios (HR) with 95% CIs will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients under 15 years of age
* Newly diagnosed with acute lymphoblastic leukemia
* Diagnosis confirmation by bone marrow aspiration and immunophenotype
* Attended in the participating Hospitals.

Exclusion Criteria:

- Patients with Down Syndrome (for being a population with different disease behavior and cytogenetic alterations than patients without this genetic condition)

Ages: 1 Day to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study variables and data will be collected from the clinical files. The information collected by the surveyors will be delivered weekly to our Research Unit, where the field work coordinators will be in charge of assigning them a folio number, reviewing the collection instrument and passing it on to the personnel in charge of capturing the information. In addition, the fieldwork coordinators will supervise the collection of information, the search for files in the archive, the capture of information and will be responsible for keeping the project's database up to date.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | year 5
  Deaths of patients occurring during the follow-up period will be collected. The cause of death and the date that this occurred will be also registered. In the case of patients alive at the end of follow-up, the date of the last visit to the hospital will be collected.
Disease-free survival | year 5
  Clinical data and by complementary examinations indicating that there is reappearance of the disease after complete remission has been achieved, presence of blasts > 5% in bone marrow (bone marrow relapse) or presence of blasts in cerebrospinal fluid fluid (CNS relapse), testicular infiltration by blasts in the biopsy (testicular relapse), combined (bone marrow/CNS) at any time during treatment . In case the patient has relapsed, the site of relapse will be collected (bone marrow, CNS, testicle, ovary, eye, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Juan M Mejía-Arangure, PhD, Principal Investigator — Instituto Mexicano del Seguro Social/Instituto Nacional de Medicina Genomica
Locations (3):
- Mexico (3):
  - Centro Médico Nacional Hospital General La Raza, IMSS, Mexico City
  - Hospital General Regional Num 1 Carlos McGregor Sánchez Navarro, IMSS, Mexico City
  - Hospital de Pediatria "Dr. Silvestre Frenk Freund" CMN Siglo XXI, IMSS, Mexico City

IPD SHARING:
Plan to Share IPD: No
The Ethics Committee asked for not making any individual participant data available

REFERENCES:
- [Result] Nunez-Enriquez JC, Gil-Hernandez AE, Jimenez-Hernandez E, Fajardo-Gutierrez A, Medina-Sanson A, Flores-Lujano J, Espinoza-Hernandez LE, Duarte-Rodriguez DA, Amador-Sanchez R, Penaloza-Gonzalez JG, Torres-Nava JR, Espinosa-Elizondo RM, Flores-Villegas LV, Merino-Pasaye LE, Perez-Saldivar ML, Dorantes-Acosta EM, Cortes-Herrera B, Solis-Labastida KA, Nunez-Villegas NN, Velazquez-Avina MM, Rangel-Lopez A, Gonzalez-Avila AI, Santillan-Juarez JD, Garcia-Velazquez AJ, Jimenez-Morales S, Bekker-Mendez VC, Rosas-Vargas H, Mata-Rocha M, Sepulveda-Robles OA, Martin-Trejo JA, Mejia-Arangure JM. Overweight and obesity as predictors of early mortality in Mexican children with acute lymphoblastic leukemia: a multicenter cohort study. BMC Cancer. 2019 Jul 18;19(1):708. doi: 10.1186/s12885-019-5878-8. PMID 31319816